CLINICAL TRIAL: NCT03325998
Title: Effect of Gait Training With a Walking Assist Robot on Gait Function and Balance in Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-04-061
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2017-10

CONDITIONS: Gait, Unsteady; Healthy
Keywords: Exoskeleton Device; Elderly; Gait rehabilitation
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait training group (Experimental): Gait training with Samsung Hip Assist v1
  All subjects receive gait training 3 times per week for 8 weeks for 24 training sessions.
  Interventions: Device: Samsung Hip Assist v1

INTERVENTIONS:
Device: Samsung Hip Assist v1 — All subjects receive gait training 3 times per week for 8 weeks for 24 training sessions. Each session is directed by a licensed physical therapist and lasted 60 min including rest period of 10 min. Brain activity and gait assessment is performed at visits 0 (baseline), 24 (post-test), and at 3 months (follow-up) after training.

SUMMARY:
The purpose of this study was to investigate the effects of gait training with the new wearable hip assist robot developed by Samsung Advance Institute of Technology (Samsung Electronics Co, Ltd, Korea) in elderly adults.

DETAILED DESCRIPTION:
Eight elderly adults will participate in this study. All subjects will receive training 3 times per week for 8 weeks for 24 training sessions. Each session is directed by a licensed physical therapist and lasted 60 min (including rest period of 10 min). Brain activity and gait assessment will be performed at visits 0 (baseline), 24 (post-test), and at 3 months (follow-up) after training.

Primary objective is to demonstrate the effects of hip assist robot on spatio-temporal parameters measured by motion capture system (Motion Analysis Corporation, Santa Rosa, CA, USA), muscle activation patterns measured by surface electromyography (sEMG) (Noraxon Inc., Scottsdale, AZ, USA), metabolic energy cost parameters measured by portable cardiopulmonary metabolic system (Cosmed K4B2, Rome, Italy) and cortical activation measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany).

Secondary objective is to demonstrate the effects of hip assist robot on motor function improvement evaluated by Short Physical Performance Battery Protocol and Score Sheet (SPPB), Berg Balance Scale (BBS), Dynamic Gait Index (DGI), Timed Up and Go (TUG) test, Push and Release (P&R) test, Functional Reach Test (FRT), Korean version Fall Efficacy Scale (K-FES), Manual Muscle Test (MMT) and Range of Motion (ROM).

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 65 and 84 years elderly adults who had no neurological or musculoskeletal abnormalities affecting gait
2. Ability to walk at least 10m regardless of assist devices
3. High levels of physical performance (SPPB > 7)
4. Subject is willing to be randomized to the control group or the treatment group

Exclusion Criteria:

1. History of any diseases (eg. lower extremity orthopedic diseases, neurologic disorders, cardiovascular disease, heart failure, uncontrolled hypertension that affect walking capacity, efficiency, and endurance)
2. Severe visual impairment or dizziness that increases the risk of falls

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test from baseline in gait speed | session 0 (initial visit); session 24 (at approximately 8 weeks); at 3 months (follow-up)
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea